CLINICAL TRIAL: NCT06922045
Title: A Phase III Clinical Study on the Efficacy and Safety of STSP-0601 for Injection in Patients With Hemophilia Associated With Inhibitors, With a Multicenter, Open Evaluation Approach
Brief Title: Phase III Clinical Trial of STSP-0601 for Injection in Hemophilia Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu BioJeTay Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STSP-0601-05
Record Dates: First submitted 2025-03-13; First posted 2025-04-10 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Continuous administration of STSP-0601 (Experimental)
  Interventions: Drug: STSP-0601 for Injection

INTERVENTIONS:
Drug: STSP-0601 for Injection — Evaluation of the Efficacy of Single-Dose and Continuous Administration of STSP-0601 Injection for the Treatment of Bleeding in Patients with Hemophilia A or B with Inhibitors

SUMMARY:
This study will assess the efficacy of multiple-dose of STSP-0601 for the treatment of bleeding episodes in hemophilia A or B patients with inhibitor

ELIGIBILITY:
Inclusion Criteria:

1. 12 ≤age≤70 years of age.
2. Hemophilia A or B patients.
3. Peak historical inhibitor titer ≥ 5 BU and a positive inhibitor test when enrolled.
4. Establish proper venous access.
5. There were at least 3 bleeding events that required treatment occurred in the past 6 months before screening.
6. Agree to use adequate contraception to avoid pregnancy.
7. Provide signed informed consent.

Exclusion Criteria:

1. Have any coagulation disorder other than hemophilia.
2. Plan to receive prophylactic treatment of coagulation factor during the trail.
3. Patients plan to receive Emicizumab during the trial.
4. Patients received anticoagulant or antifibrinolytic therapy 7 days before the first administration or plan to receive these drugs during the trial.
5. Have a history of arterial and/or venous thrombotic events.
6. Platelet <100×109/L.
7. Hemoglobin<90g/L.
8. Severe liver or kidney disease.
9. Severe bleeding event occurred within 4 weeks before the first administration.
10. Accepted major operation or blood transfusion within 4 weeks before the first administration.
11. Have a known allergy to STSP-0601.
12. Pregnant, lactating, or blood pregnancy test positive female subjects
13. Participate in other clinical research within 4 weeks before enrollment (except for participating in prothrombin complex, FVII, FVIIa, FVIII, FIX trails).
14. Within 1 day before the first administration, FVII, FVIIa, tranexamic acid, and aminocaproic acid were used. Within 3 days before the first administration, prothrombin complex, FVIII, and FIX were used. Within 4 weeks, treatment with Emicizumab was received.
15. Patients not suitable for the trail according to the judgment of the investigators.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
12 hours effective hemostasis rate | 12 hours after the first administration

SECONDARY OUTCOMES:
Effective hemostasis rate at the first 12 hours bleeding visit | 12 hours after the first administration
12 hours excellent + good rate | 12 hours after the first administration
The number of medication required for effective hemostasis within 12 hours | 12 hours after the first administration
The amount of medication (U/kg) required for effective hemostasis within 12 hours | 12 hours after the first administration
8-hours effective hemostasis rate | 8 hours after the first administration
8-hours excellent + good rate | 8 hours after the first administration
Complete + significant relief rate | 4 hours, 8 hours, 12 hours, 24 hours after the first administration
The time to achieve complete/significant remission after the first administration | From the time after the first administration until within 72 hours after the last administration
Rescue treatment rate | Within 72 hours after the last administration
The time from the onset of bleeding to complete/significant relief | Within 72 hours after the last administration
The effective hemostasis rate of the target joint | From 12 hours after the first administration to 72 hours after the last administration

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, Ph.D, Principal Investigator — Hospital of Hematology, Chinese Academy of Medical Sciences
Locations (18):
- China (18):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Lanzhou University First Hospital, Lanzhou, Gansu
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - The First affiliated hospital of Guangxi Medical University, Nanning, Guangxi
  - North China University of Science and Technology Affiliated Hospital, Tangshan, Hebei
  - Harbin First Hospital Hematology Tumor Research Center, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Huazhong University of Science and Technology Union Hospital, Wuhan, Hubei
  - Jiangsu Provincial Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jinan Central Clinical College of Shandong First Medical University, Jinan, Shandong
  - Second hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Xi'an Central Hospital, Xi’an, Shanxi
  - Sichuan Academy of Medical Sciences＆Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Hospital of Hematology, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Wenzhou People's Hospital, Wenzhou, Zhejiang